CLINICAL TRIAL: NCT05350696
Title: Comparative Study Between Erector Spinae Plane Block Versus Intravenous Morphine as Postoperative Analgesia After Spine Surgeries .
Brief Title: Comparative Study Between ESPB Versus IV Morphine as Postoperative Analgesia After Spine Surgeries .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Aboelhamed Abdelrahman, resident doctor at Anasthesia department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Soh-Med-22-03-10
Record Dates: First submitted 2022-03-15; First posted 2022-04-28 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Discectomy; Vertebral Fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane block group (Active Comparator): (30 patients) will receive bilateral ultrasound guided erector spinae plane block using plain bupivacaine 100 mg diluted to volume using normal saline to achieve 50% concentration ( 50 mg plain pubivicaine in each side ).
  Interventions: Drug: Erector Spinae plane block (plain pubivicaine)
- Intravenous Morphine group (Active Comparator): (30 patients) will receive 0.1 mg /kg of intravenous morphine diluted to 10 ml volume using saline at the end of the operation.
  Interventions: Drug: Intravenous morphine group

INTERVENTIONS:
Drug: Erector Spinae plane block (plain pubivicaine) — The erector spinae block is achieved by injecting the local anesthetic solution (with possible adjuvants) between the erector spinae muscles (iliocostalis, longissimus, spinalis/ from lateral to medial) and the transverse process .
  The technique is performed under ultrasound guidance.
  Other Names: ESPB group
  Arms: Erector Spinae Plane block group
Drug: Intravenous morphine group — patients will receive 0.1 mg /kg of intravenous morphine diluted to 10 ml volume using saline at the end of the operation.
  Other Names: Morphine group
  Arms: Intravenous Morphine group

SUMMARY:
Postoperative pain is often severe in patients undergoing lumbar surgery. Due to postoperative pain, patients are unwilling to get out of bed at an early stage, which affects their recovery.

Erector spinae plane block (ESPB) as a new trunk fascia block technique was proposed in 2016. ESPB has aroused the interest of many nerve block experts. The benefits of ESPB are not yet demonstrated. The specific mechanism is still controversial.

The erector spinae block is achieved by injecting the local anesthetic solution (with possible adjuvants) between the erector spinae muscles (iliocostalis, longissimus, spinalis/ from lateral to medial) and the transverse process .

The technique is performed under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar Disc Prolapse.
* Fracture Lumbar Vertebrae

Exclusion Criteria:

1. Patient refusal.
2. Drug abuse.
3. Patient with significant neurological, psychiatric or neuromuscular disease.
4. Chronic pain on medicine.
5. known allergy to the study medications.
6. Infection at the site of infiltration.
7. Patients with bleeding tendency.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia . | 24 hours after surgery
  The study will include 60 adult patients undergoing uncomplicated spine surgery under general anesthesia.
  At the end of operation , Patients will be randomly divided using closed enveloped method into two equal groups.
  * Group 1, (30 patients) will receive bilateral ultrasound guided erector spinae plane block using plain bupivacaine 100 mg diluted to volume using normal saline to achieve 50% concentration ( 50 mg plain pubivicaine in each side ).
  * Group 2, (30 patients) will receive 0.1 mg /kg of intravenous morphine diluted to 10 ml volume using saline at the end of the operation.
  postoperative pain assessment according to visual analogue scale ( VAS ) within 24 hours after the surgery.
  0 - 3 mild pain ( better outcome )
  4 - 6 moderate pain
  7 - 10 severe pain
  > 10 unbearable pain ( worst outcome)

SECONDARY OUTCOMES:
Avoid side effects of using systemic morphine. | 24 hours after surgery
  use of intravenous morphine is mostly followed by undesirable side effects such as postoperative nausea and vomiting,urine retention and constipation.
  so the target of this study is to show that if ESPB is more preferrable to IV morphine as regard both : postoperative anagesia and avoidance of side effects of systemic morphine.
  patients of morphine group will be asked about having nausea or vomiting after surgery and over 24 hours after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth. 2017 Mar 1;118(3):474-475. doi: 10.1093/bja/aex013. No abstract available. PMID 28203765
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Melvin JP, Schrot RJ, Chu GM, Chin KJ. Low thoracic erector spinae plane block for perioperative analgesia in lumbosacral spine surgery: a case series. Can J Anaesth. 2018 Sep;65(9):1057-1065. doi: 10.1007/s12630-018-1145-8. Epub 2018 Apr 27. PMID 29704223
- [Background] Tseng V, Xu JL. Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: Is There a Better Option? J Neurosurg Anesthesiol. 2021 Jan;33(1):92. doi: 10.1097/ANA.0000000000000631. No abstract available. PMID 31343504